CLINICAL TRIAL: NCT03806179
Title: A Phase 1b Open-label Study of Betalutin in Combination With Rituximab in Patients With Relapsed/Refractory Follicular Lymphoma (Archer-1)
Brief Title: Study of Safety and Efficacy of Betalutin and Rituximab in Patients With FL
Acronym: LYMRIT-37-07
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nordic Nanovector (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LYMRIT -37-07(Archer-1); 2017-004506-18 (Other: EudraCT)
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Non Hodgkin Lymphoma; Follicular Lymphoma; Relapsed Follicular Lymphoma
Keywords: Radioimmunotherapy; Lu-177; Betalutin; Phase 1b; Combination; Rituximab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 MBq/kg Betalutin with rituximab treatment (Experimental): 10 MBq/kg Betalutin administered with lilotomab pre-dose on day 0; rituximab administered weekly x 4 doses from day 7, then every 3 months for 2 years
  Interventions: Drug: 10 MBq/kg Betalutin
- 15 MBq/kg Betalutin with rituximab treatment (Experimental): 15 MBq/kg Betalutin administered with lilotomab pre-dose on day 0; rituximab administered weekly x 4 doses from day 7, then every 3 months for 2 years
  Interventions: Drug: 15 MBq/kg Betalutin

INTERVENTIONS:
Drug: 10 MBq/kg Betalutin — 10 MBq/kg Betalutin, lilotomab 40mg, rituximab 375 mg/m2
  Arms: 10 MBq/kg Betalutin with rituximab treatment
Drug: 15 MBq/kg Betalutin — 15 MBq/kg Betalutin, lilotomab 40mg, rituximab 375 mg/m2
  Arms: 15 MBq/kg Betalutin with rituximab treatment

SUMMARY:
This study is a Phase 1b, open-label, single arm dose escalation study of Betalutin followed by rituximab in patients with previously treated follicular lymphoma. The purpose of this study is to characterise the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary anti-tumour activity of Betalutin in combination with rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥18 years at the time of signing the informed consent
* ECOG performance status of 0-2
* Histologically confirmed diagnosis (by 2008 World Health Organization [WHO] classification) of follicular lymphoma (grade 1, 2 or 3a)
* At least one (but not more than 3) prior regimens with an anti-CD20 antibody (alone or in combination with chemotherapy), with documented relapsed, refractory disease (must not be anti-CD20 antibody-refractory) or PD
* Presence of at least one bi-dimensionally measurable lesion by CT or MRI: longest diameter (LDi) >1.5 cm for a nodal lesion; LDi >1.0 cm for an extranodal lesion within 28 days prior to start of treatment
* Normal organ and bone marrow function defined as:

  1. Absolute neutrophil count ≥1.5 x 109/L;
  2. Platelet count ≥150 x 109/L;
  3. Haemoglobin ≥9 g/dL;
  4. Total bilirubin ≤1.5 x upper limit of normal (ULN) (except patients with documented Gilbert's syndrome [<3.0 mg/dL]);
  5. Aspartate transaminase (AST); Alanine transaminase (ALT) or Alkaline phosphatase (ALP) ≤2.5 x ULN (or ≤5.0 x ULN if liver involvement by primary disease);
  6. Adequate renal function as demonstrated by a serum creatinine within the upper limit of normal range
* Bone marrow involvement by lymphoma <25%
* Life expectancy >3 months
* Negative hepatitis B, hepatitis C and human immunodeficiency virus (HIV) screening tests
* Patients must agree to use effective contraception for 12 months following last study drug administration

Exclusion criteria:

* Previous haematopoietic stem cell transplantation (autologous and allogenic)
* Evidence of histological transformation from FL to DLBCL at time of screening.
* Previous total body irradiation
* Chemotherapy, immunotherapy or investigational therapy within 28 days before the start of study drug administration (corticosteroid treatment at doses of ≤20 mg/day, topical or inhaled corticosteroids, granulocyte colony-stimulating factor [G-CSF] or granulocyte-macrophage colony-stimulating factor [GM CSF] are permitted up to 2 weeks prior to start of study treatment) or failure to recover from AEs associated with prior treatment
* Previous treatment with radioimmunotherapy
* Patients who are receiving any other investigational medicinal products
* Known or suspected central nervous system (CNS) involvement of lymphoma
* History of a previous treated cancer except for the following:

  1. adequately treated local basal cell or squamous cell carcinoma of the skin
  2. cervical carcinoma in situ
  3. superficial bladder cancer or localised prostate cancer undergoing surveillance or surgery
  4. localised breast cancer treated with surgery and radiotherapy but not including systemic chemotherapy
  5. other adequately treated Stage 1 or 2 cancer currently in CR
* Pregnant or lactating women
* Exposure to another CD37 targeting drug
* A known hypersensitivity to RTX, lilotomab, Betalutin or murine proteins or any excipient used in RTX, lilotomab or Betalutin
* Receipt of live, attenuated vaccine within 30 days prior to enrolment
* Evidence of severe or uncontrolled systemic diseases (e.g. ongoing infection, respiratory, cardiac, hepatic or psychiatric conditions) which in the Investigator's opinion would compromise the protocol objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fosså, MD.PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Klinika Hematoonkologie, Ostrava, Porubá, Czechia
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Repetto-Llamazares AHV, Malenge MM, O'Shea A, Eiriksdottir B, Stokke T, Larsen RH, Dahle J. Combination of 177 Lu-lilotomab with rituximab significantly improves the therapeutic outcome in preclinical models of non-Hodgkin's lymphoma. Eur J Haematol. 2018 Oct;101(4):522-531. doi: 10.1111/ejh.13139. Epub 2018 Aug 31. PMID 29993152
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 10 MBq/kg Betalutin With Rituximab Treatment | 15 MBq/kg Betalutin With Rituximab Treatment
Started | 4 (Includes one participant who received 10 MBq/kg instead of 15 MBq/kg in error) | 3
Completed | 4 | 1
Not Completed | 0 | 2
Not completed — Progressive disease | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 MBq/kg Betalutin With Rituximab Treatment | 15 MBq/kg Betalutin With Rituximab Treatment | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Norway | 4 | 2 | 6
  Czechia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability: Frequency and Severity of Adverse Events (CTCAE v4.03)
Description: Safety and tolerability of Betalutin in combination with rituximab as determined by the frequency and severity of adverse events (CTCAE v4.03) in the first 12 weeks after Betalutin
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 10 MBq/kg Betalutin With Rituximab Treatment | 15 MBq/kg Betalutin With Rituximab Treatment
Number analyzed (Participants) | 4 | 3
Participants
  Number of participants with dose limiting toxicities in the first 12 weeks | 0 | 0
  Number of participants with adverse events in the first 12 weeks | 3 | 3
  Number of participants with SAEs in the first 12 weeks | 0 | 0
  Number of participants with Betalutin related adverse events in the first 12 weeks | 1 | 3
  Number of participants with CTCAE Grade 3 or 4 adverse events in the first 12 weeks | 2 | 2

2. Secondary Outcome: Preliminary Anti-tumour Activity
Description: Best overall response of combination treatment using tumour responses based on CT and PET/CT imaging (classified as as complete response, partial response, no response/stable disease or progressive disease as described in "Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification")
Time Frame: 25 months
Measure: Count of Participants; unit: Participants
Arm/Group | 10 MBq/kg Betalutin With Rituximab Treatment | 15 MBq/kg Betalutin With Rituximab Treatment
Number analyzed (Participants) | 4 | 3
Participants
  Complete response | 3 | 2
  Partial response | 1 | 1

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from the time of informed consent until 4 weeks after the last rituximab dose, up to 25 months. Thereafter treatment related AEs were collected up to 36 months for the first two participants only.
Description: Treatment emergent AEs from the first dose of rituximab are presented. Under protocol Versions 1 to 3, it was planned to collect treatment-related AEs for the duration of the follow-up period, up to 5 years. This period was removed under protocol Version 4; only the first two participants had entered the follow-up period at the time this version was approved, therefore only these two participants had treatment-related AEs collected up to 36 months before follow-up was closed.
Arm/Group | 10 MBq/kg Betalutin With Rituximab Treatment | 15 MBq/kg Betalutin With Rituximab Treatment
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 MBq/kg Betalutin With Rituximab Treatment (N=4) | 15 MBq/kg Betalutin With Rituximab Treatment (N=3)
Erysipelas (Infections and infestations) | 1 | 0 — Occurred >92 days (12 weeks) after Betalutin injection
Fall (Injury, poisoning and procedural complications) | 1 | 0 — Occurred >92 days (12 weeks) after Betalutin injection
Bronchitis viral (Infections and infestations) | 1 | 0 — Occurred >92 days (12 weeks) after Betalutin injection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 MBq/kg Betalutin With Rituximab Treatment (N=4) | 15 MBq/kg Betalutin With Rituximab Treatment (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Facial pain (General disorders) | 0 | 1
Influenza-like illness (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 1
Restless leg syndrome (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Primary progressive aphasia (Nervous system disorders) | 1 | 0
Nerve degeneration (Nervous system disorders) | 1 | 0
Axillary pain (General disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling (General disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Post-traumatic headache (Nervous system disorders) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Whilst the protocol makes reference to a separate statistical analysis plan, given that only seven participants were enrolled and the originally planned expansion phase in a further 20-25 participants was not performed (removed under protocol Version 4.0) a separate detailed statistical analysis plan was not generated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT03806179/Prot_SAP_000.pdf